CLINICAL TRIAL: NCT06935370
Title: EASi-HF Reduced - A Phase III Double-blind, Randomised, Parallel-group Superiority Trial to Evaluate Efficacy and Safety of the Combined Use of Oral Vicadrostat (BI 690517) and Empagliflozin Compared With Placebo and Empagliflozin in Participants With Symptomatic Chronic Heart Failure (HF: NYHA II-IV) and Left Ventricular Ejection Fraction (LVEF) < 40%
Brief Title: A Study to Test Whether Vicadrostat (BI 690517) in Combination With Empagliflozin Helps People With Heart Failure and a Weak Pumping Function of the Left Side of the Heart
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1378-0018; 2024-519525-38-00 (EU CTIS Number); U1111-1317-0692 (Other: WHO - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-04-17; First posted 2025-04-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- vicadrostat/empagliflozin treatment group (Experimental)
  Interventions: Drug: vicadrostat; Drug: empagliflozin
- Placebo to vicadrostat/empagliflozin treatment group (Placebo Comparator)
  Interventions: Drug: empagliflozin; Drug: Placebo

INTERVENTIONS:
Drug: vicadrostat — vicadrostat
  Arms: vicadrostat/empagliflozin treatment group
Drug: empagliflozin — empagliflozin
Drug: Placebo — Placebo matching vicadrostat
  Arms: Placebo to vicadrostat/empagliflozin treatment group

SUMMARY:
This study is open to adults with chronic heart failure (HF) who have a reduced left ventricular ejection fraction (LVEF) of less than 40%. People can join the study if they have been diagnosed with chronic HF at least 3 months before the study. The purpose of this study is to find out whether a medicine called vicadrostat, in combination with another medicine called empagliflozin, helps people with chronic heart failure.

In this study, participants are put into 2 groups randomly. Participants have an equal chance of being in either group. One group takes vicadrostat/empagliflozin tablets, and the other group takes placebo/empagliflozin tablets. Placebo tablets look like vicadrostat tablets but do not contain any medicine. Participants take the study medicines as tablets once a day for between 1 and about 3.5 years. During this time, they can continue their regular treatment for heart failure.

Participants can stay in the study as long as they benefit from treatment and can tolerate it, for a maximum of about 3.5 years. During this time, they visit the study site regularly. The exact number of visits is different for each participant, depending on how long they stay in the study. The study staff may also contact the participants by phone. Participants also regularly answer questions about their well-being. The doctors document when participants experience worsening of their heart failure symptoms, must go to hospital due to heart failure, or die during the study. The time until these events are observed is compared between the treatment groups to see whether the treatment works. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria:

1. At least 18 years old and at least at the legal age of consent in countries where it is greater than 18 years
2. Signed and dated written informed consent in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
3. Male or female participants. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria and instructions on the duration of their use is provided in the protocol.
4. Chronic heart failure (HF) diagnosed at least 3 months before Visit 1, and in New York Heart Association (NYHA) classes II to IV at Visit 1, with left ventricular ejection fraction (LVEF) < 40% per local reading (obtained by echocardiography, radionuclide ventriculography, invasive angiography, magnetic resonance imaging (MRI), or computed tomography (CT)).
5. Elevated N-terminal pro-brain natriuretic peptide (NT-proBNP) at Visit 1, analysed at the central laboratory
6. Treated according to best possible standard of care (SOC) (disregarding sodium-dependent glucose co-transporter 2 inhibitor (SGLT2i) and mineralocorticoid receptor antagonist (MRA)) in accordance with applicable heart failure (HF) local/international guidelines and judgement of the investigator.

Additional inclusion criteria apply.

Exclusion criteria:

1. Treatment with an MRA (e.g. spironolactone, eplerenone, finerenone) within 14 days prior to Visit 1 or requiring such treatment before randomisation or planned during the trial based on the judgment of the investigator. Treatment with an MRA should not be discontinued with the intention of study enrolment.
2. Treatment with amiloride or other potassium-sparing diuretic within 14 days prior to Visit 1 or requiring such treatment before randomisation or planned during the trial based on the judgment of the investigator.
3. Receiving the following treatments:

   * A direct renin inhibitor (e.g. aliskiren) at Visit 2
   * More than one angiotensin-converting enzyme inhibitor (ACEi), angiotensin receptor blocker (ARB) or angiotensin receptor-neprilysin inhibitor (ARNi) used simultaneously at Visit 2
   * Other aldosterone synthase inhibitors, e.g. baxdrostat at Visit 2 or planned during the trial
   * Systemic mineralocorticoid replacement therapy (e.g. fludrocortisone) at Visit 2
   * In case of acute decompensated HF:

     * i.v. inotrope, i.v. vasodilating drug (e.g. nitrate, nitroprusside), or i.v. natriuretic peptide (e.g. nesiritide, carperitide), or mechanical support (e.g. intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, any ventricular assist device) within 24 hours prior to randomisation
     * i.v. diuretic with a dose that has been increased/intensified within 6 hours prior to randomisation (a stable dose of an i.v. diuretic is not exclusionary)
4. Myocardial infarction (MI), transient ischemic attack (TIA), stroke, coronary artery bypass graft surgery (CABG), heart valve surgery/intervention or any other major surgery (major according to the investigator's assessment) within 90 days prior to Visit 2, or scheduled for major elective surgery (e.g. hip replacement, CABG)
5. Percutaneous coronary intervention (PCI) or any angiography using iodinated contrast agents in the 7 days prior to Visit 2
6. Heart transplant recipient, awaiting heart transplant, or currently implanted left ventricular assist device (LVAD)
7. Known cardiomyopathy based on infiltrative diseases (e.g. amyloidosis), accumulation diseases (e.g. haemochromatosis, Fabry disease), muscular dystrophies, hypertrophic obstructive cardiomyopathy or known pericardial constriction, or cardiomyopathy with potentially reversible cause such as stress or peripartum cardiomyopathy or cardiomyopathy induced by chemotherapy within 12 months prior to Visit 1 and until Visit 2
8. Acute inflammatory heart disease, such as acute myocarditis, within 90 days preceding prior to Visit 1 and until Visit 2 Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4200 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2029-02-04 (Estimated); Study Completion 2029-02-22 (Estimated)

PRIMARY OUTCOMES:
Time to first event of Cardiovascular (CV) death, or Hospitalisation for heart failure (HHF), or Urgent heart failure (HF) visit | up to 43 months

SECONDARY OUTCOMES:
Key secondary endpoint: Time to first event of cardiovascular death or hospitalisation for heart failure | up to 43 months
Key secondary endpoint: Occurrences of hospitalisation for heart failure (first and recurrent) | up to 43 months
Key secondary endpoint: Absolute change from baseline in Kansas City Cardiomyopathy Questionnaire-Total Symptom Score (KCCQ-TSS) at Week 32 | at baseline, at week 32
  The KCCQ is a participant reported outcome. The KCCQ is a 23-item self-administered questionnaire designed to evaluate physical limitations, symptoms (frequency, severity, and changes over time), social limitations, self-efficacy, and quality of life in people with heart failure.
  The symptom frequency and symptom burden domains are merged into a total symptom score (TSS).
  Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Key secondary endpoint: Time to cardiovascular death | up to 43 months
Key secondary endpoint: Time to all-cause mortality | up to 43 months
Time to first hospitalisation for heart failure | up to 43 months
Time to first occurrence of death from kidney failure, chronic dialysis* or renal transplant or onset of sustained reduction of ≥ 50% estimated glomerular filtration rate (eGFR) or onset of sustained eGFR (CKD-EPI)cr < 10 mL/min/1.73 m² | from baseline, up to 43 months
  * Chronic dialysis is defined as dialysis continuing for at least 30 days. For this composite renal endpoint the Chronic Kidney Disease Epidemiology Collaboration creatinine ((CKD-EPI)cr) equation is used.
Absolute change from baseline in Kansas City Cardiomyopathy Questionnaire- Clinical Summary Score (KCCQ-CSS) at Week 32 | at baseline, at week 32
  The KCCQ is a participant reported outcome. The KCCQ is a 23-item self-administered questionnaire designed to evaluate physical limitations, symptoms (frequency, severity, and changes over time), social limitations, self-efficacy, and quality of life in people with heart failure.
  The Clinical Summary Score (CSS) of the KCCQ provides a measure of symptoms and physical limitations associated with heart failure.
  Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Absolute change from baseline in Kansas City Cardiomyopathy Questionnaire-Total Symptom Score (KCCQ-TSS) at Week 52 | at baseline, at week 52
  The KCCQ is a participant reported outcome. The KCCQ is a 23-item self-administered questionnaire designed to evaluate physical limitations, symptoms (frequency, severity, and changes over time), social limitations, self-efficacy, and quality of life in people with heart failure.
  The symptom frequency and symptom burden domains are merged into a total symptom score (TSS).
  Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Absolute change from baseline in Kansas City Cardiomyopathy Questionnaire- Overall Summary Score (KCCQ-OSS) at Week 32 | at baseline, at week 32
  The KCCQ is a participant reported outcome. The KCCQ is a 23-item self-administered questionnaire designed to evaluate physical limitations, symptoms (frequency, severity, and changes over time), social limitations, self-efficacy, and quality of life in people with heart failure.
  In the KCCQ, an overall summary score (OSS) can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains.
  Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Absolute change from baseline in KCCQ-OSS at Week 52 | at baseline, at week 52
  The KCCQ is a participant reported outcome. The KCCQ is a 23-item self-administered questionnaire designed to evaluate physical limitations, symptoms (frequency, severity, and changes over time), social limitations, self-efficacy, and quality of life in people with heart failure.
  In the KCCQ, an overall summary score (OSS) can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains.
  Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Absolute change from baseline in systolic blood pressure (SBP) [mmHg] at Week 32 in participants with baseline SBP ≥ 130 mmHg | at baseline, at week 32
Absolute change from baseline in diastolic blood pressure (DBP) [mmHg] at Week 32 in participants with baseline DBP ≥ 80 mmHg | at baseline, at week 32

CONTACTS AND LOCATIONS:
Locations (634):
- United States (107):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Drug Research and Analysis Corporation, Montgomery, Alabama
  - Cure Clinical Research, Beverly Hills, California
  - Valley Clinical Trials, Inc., Covina, California
  - North Coast Cardiology, Encinitas, California
  - Orange County Research Center, Lake Forest, California
  - Merced Vein and Vascular Center, Merced, California
  - Radin Cardiovascular Medical Group, Newport Beach, California
  - Amicis Research Center, Northridge, California
  - University of California San Diego, San Diego, California
  - Paradigm Clinical Research - San Diego, San Diego, California
  - Care Access Research, Thousand Oaks, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Bay Area Cardiology, Brandon, Florida
  - Cardiology Associates Research Co., Daytona Beach, Florida
  - Suncoast Research Associates, LLC, Doral, Florida
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - Velocity Clinical Research-Hallandale Beach-67888, Hallandale, Florida
  - University of Florida, Jacksonville, Florida
  - East Coast Institute For Research, LLC, Jacksonville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Central Therapy Center, Inc., Miami, Florida
  - Inpatient Research Clinic, LLC, Miami Lakes, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - St. Johns Center for Clinical Research, Saint Augustine, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Cozy Research LLC, Wesley Chapel, Florida
  - Clinical Site Partners, LLC, Winter Park, Florida
  - Atlanta Clinical Research Centers, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - NSC Research Inc, Johns Creek, Georgia
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Illinois Masonic Hospital, Chicago, Illinois
  - Chicago Medical Research, Hazel Crest, Illinois
  - Clinical Investigation Specialists, Inc., Libertyville, Illinois
  - AMR Park Ridge, Park Ridge, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Midwest Cardiovascular Research and Education Foundation, Elkhart, Indiana
  - St. Francis Medical Group-Indiana Heart Physicians, Inc, Indianapolis, Indiana
  - Indiana Medical Research Institute, Merrillville, Indiana
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - Reid Hospital, Richmond, Indiana
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kansas Nephrology Research Institute, LLC, Wichita, Kansas
  - Robert J Dole Veterans Affairs Medical Center, Wichita, Kansas
  - West Houston Area Clinical Trial Consultants, LLC, Wichita, Kansas
  - Norton Healtcare - Norton Heart and Vascular Institute, Louisville, Kentucky
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Grace Research, LLC-Shreveport-64616, Shreveport, Louisiana
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants, Beltsville, Maryland
  - Capitol Cardiology Associates, Lanham, Maryland
  - McLaren Bay Region Medical Center, Bay City, Michigan
  - Cardiology and Vascular Associates - CAVA, Bloomfield Hills, Michigan
  - Michigan Healthcare Professionals Pulse Cardiology, Farmington Hills, Michigan
  - St. John Providence Hospital, Novi, Michigan
  - Michigan Heart, PC, Ypsilanti, Michigan
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Jackson Heart Clinic, P.A., Jackson, Mississippi
  - North Kansas City Hospital, Kansas City, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - St. Louis Heart and Vascular, P.C., St Louis, Missouri
  - Be Well Clinical Studies, Omaha, Nebraska
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - Garden State Heart Care, PC, Manalapan, New Jersey
  - Bassett Medical Center, Cooperstown, New York
  - Mount Sinai Hospital-New York-52529, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - IMA Clinical Research Lenoir, Lenoir, North Carolina
  - Pinehurst Medical Clinic, Inc. - East, Pinehurst, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Piedmont Healthcare, Inc., Statesville, North Carolina
  - Wilmington Health, Wilmington, North Carolina
  - VA Northeast Ohio Healthcare System, Cleveland, Ohio
  - K and R Research LLC, Marion, Ohio
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Bon Secours Medical Group Greenville Specialty Care, LLC, Greenville, South Carolina
  - Monument Health, Rapid City, South Dakota
  - Pharmatex Research, Amarillo, Texas
  - Amarillo Heart Clinical Research Institute, Incorporated, Amarillo, Texas
  - NextStage Clinical Research, Beaumont, Texas
  - Headlands Research Brownsville, Brownsville, Texas
  - Texas Health Research and Education Institute, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Helios CR Inc - Fort Worth, Fort Worth, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - DM Clinical Research Dallas, Irving, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - North Texas Research Associates, McKinney, Texas
  - Texas Institute Of Cardiology, McKinney, Texas
  - Stryde Research, Plano, Texas
  - Accurate Clinical Research, Inc., Richmond, Texas
  - Revival Research Institute, LLC., Sherman, Texas
  - Baylor Scott and White Health, Temple, Texas
  - Northwest Heart Center, Tomball, Texas
  - NextStage Clinical Research, Waco, Texas
  - Virginia Heart - Falls Church, Falls Church, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Carilion Clinic, Roanoke, Virginia
- Argentina (39):
  - Inst de Inv Clinicas-Bahia Blanca, Bahía Blanca
  - Hospital Regional de Bahia Blanca, Bahía Blanca
  - CIPREC, Buenos Aires
  - Centro de Investigaciones Metabolicas (CINME)-C.A.B.A-61553, C.a.b.a
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Fundacion Favaloro, Ciudad Autonoma Buenos Aires
  - Mautalen- Salud e Investigacion, Ciudad Autonoma Buenos Aires
  - Centro Medico Dra Laura Maffei, Ciudad Autonoma Buenos Aires
  - Glenny Corp. S.A. Bioclinica Argentina, Ciudad Autonoma Buenos Aires
  - Clinica Coronel Suárez, Coronel Suárez
  - Sanatorio Allende, Córdoba
  - Sanatorio Privado Duarte Quiros De Clinica Colombo SA, Córdoba
  - Well Medica, Córdoba
  - Instituto Médico DAMIC S.R.L., Córdoba
  - Centro Medico Luquez, Córdoba
  - Hospital Italiano de La Plata, La Plata
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata
  - Hospital Universitario Austral, Pilar
  - Instituto Medico CER, Quilmes
  - Instituto de Investigaciones Clínicas de Quilmes, Quilmes
  - DIM Clinica Privada, Ramos Mejía
  - INECO Neurociencias Oroño, Rosario
  - Instituto de Investigaciones Clinicas de Rosario, Rosario
  - Instituto Medico Fundacion Grupo Colaborativo Rosario Investigacion y Prevencion Medica, Rosario
  - Sanatorio Parque S.A., Rosario
  - Instituto CAICI, Rosario
  - Investigaciones Clinicas Salta (ICSAL), Salta
  - Centro Cardiovascular Salta, Salta
  - Corporacion Medica de Gral. San Martin S.A., San Martín
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán
  - Centro Integral de Arritmias Tucuman, San Miguel de Tucumán
  - Centro Modelo de Cardiologia, San Miguel de Tucumán
  - Clinica Mayo, San Miguel de Tucumán
  - Instituto de Investigaciones Clinicas San Nicolas, San Nicolás
  - Centro de Investigaciones Clinicas Baigorria, Santa Fe
  - Hospital "Dr. José Maria Cullen", Santa Fe
  - Centro de Investigaciones Clínicas del Litoral, Santa Fe
  - CEMEDIC - Centro de Especialidades Medicas, Villa Luro
- Belgium (7):
  - AZ Sint-Blasius, Dendermonde
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Sint-Lucas, Ghent
  - Grand Hôpital de Charleroi, Gilly
  - AZ Groeninge, Kortrijk
  - C.H.U. de Tivoli, La Louvière
  - CHR de la Citadelle, Liège
- Brazil (39):
  - Hospital Sirio Libanes, Bela Vista
  - Hospital Felicio Rocho, Belo Horizonte
  - Cardresearch Cardiologia Assistencial e de Pesquisas Ltda, Belo Horizonte
  - L2IP -Instituto de Pesquisas Clínicas Ltda., Brasília
  - Hospital DF Star, Brasília
  - CECAP - Centro de Cardiologia Clínica, Brasília
  - Hospital Angelina Caron, Campina Grande do Sul
  - IPECC - Instituto de Pesquisa Clínica de Campinas, Campinas
  - Hospital PUC-Campinas, Campinas
  - I9 Pesquisas Clinicas - Loema Instituto de Pesquisa Clínica e Consultores SS Ltda, Campinas
  - Hospital do Rocio, Campo Largo
  - Fundacao Universidade de Caxias do Sul, Caxias do Sul
  - PUC Trials - Núcleo de Pesquisa Clínica da Escola de Medicina da PUC-PR, Curitiba
  - Via Medica, Goiânia
  - HC-UFG - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia
  - ICM - Instituto do Coracao de Marilia, Marília
  - Hospital Vera Cruz, Minas Gerais
  - Instituto Atena de Pesquisa Clinica, Natal
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Nucleo de Pesquisa Clinica do Rio Grande do Sul (NPCRS), Porto Alegre
  - Hospital Mae de Deus, Porto Alegre
  - Hospital Esperança Recife, Recife
  - Clinicor Clínica Cardiológica LTDA/ Cardio Prime - CAPED, Ribeirão Preto
  - Instituto Brasil de Pesquisa Clinica (IBPClin), Rio de Janeiro
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - Instituto D'Or Pesquisa e Ensino - Rio de Janeiro, Rio de Janeiro
  - Hospital Cardio Pulmonar, Salvador
  - Pesquisare, Santo André
  - Praxis Pesquisa Medica, Santo André
  - Instituto Domingo Braile, São José do Rio Preto
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - CIPES - Centro Internacional de Pesquisa Clínica, São José dos Campos
  - Cpquali Pesquisa Clinica Ltda, São Paulo
  - Centro de Pesquisa Clinica - CPCLIN, São Paulo
  - CEPIC - Centro Paulista de Investigacao Clinica, São Paulo
  - Eurolatino Pesquisas Médicas Ltda., Uberlândia
  - CEDOES - Diagnóstico e Pesquisa,Vitória, Vitória
- Bulgaria (38):
  - Medical center 4LIFE Ltd., Burgas
  - MHAT Heart and brain, Burgas
  - Medical Center Doktor Staykov Ltd., Burgas
  - Diamedical Medical Center 2013, Dimitrovgrad
  - MHAT "Sveta Ekaterina-Dimitrovgrad", EOOD, Dimitrovgrad
  - Medical Center New Polyclinic Gabrovo Ltd., Gabrovo
  - MHAT Ivan Skenderov EOOD, Gotse Delchev
  - Medical Center Rodopimed EOOD, Kardzhali
  - Medical Center Hera - Kyustendil EOOD, Kyustendil
  - Tonus 2013 Ltd., Pazardzhik
  - Ambulatory Individual Practice for Cardiology Specialized Medical Care, Pernik
  - Medical Center Medconsult Pleven OOD, Pleven
  - MHAT Heart and brain, Pleven
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - MBAL Sveta Karidad EAD, Plovdiv
  - Medical Center Rusemed EOOD, Rousse
  - National Multiprofile Transport Hospital "Tzar Boris III", Sofia
  - Medical Center For Specialized Medical Help In Cardiovascular Diseases OOD, Sofia
  - University Hospital Lozenetz, Sofia
  - Alexandrovska University Hospital, Sofia
  - Diagnostic Consultative Center Alexandrovska, Sofia
  - University Multidisciplinary Hospital for Active Treatment Sveta Ekaterina EAD, Sofia
  - Medical Center Hera EOOD, Sofia
  - UMHAT "Tsaritsa Yoanna-ISUL" EAD, Sofia
  - ASOMHIDC - Individual practice "Cardio Tonus" EOOD, Sofia
  - Multiprofile Hospital MHATEM 'Pirogov', Sofia, Sofia
  - Diagnostic Consultation Center XX-Sofia EOOD, Sofia
  - MHAT "St. Sofia", Sofia
  - Kalimat Medical Center Ltd., Sofia
  - Medical Center Intermedica Ltd., Sofia
  - Medical Center Medicabilis Ltd., Sofia
  - Medical center DEA Medicals Ltd., Sofia
  - Medical Center Zara-Med EOOD, Stara Zagora
  - UMHAT Prof. Dr. Stoyan Kirkovich AD, Stara Zagora
  - MDHAT 'Dr. Stefan Cherkezov', AD, Veliko Tarnovo
  - Medical Center Medica Plus Ltd., Veliko Tarnovo
  - Medical Centre Nevromedics EOOD, Veliko Tarnovo
  - MHAT St Panteleimon, Yambol
- Canada (17):
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Saul Vizel Medicine Professional Corporation, Cambridge, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Premier Clinical Trial Network, Hamilton, Ontario
  - Elevate Clinical Research - KMH Hamilton, Kitchener, Ontario
  - KMH Cardiology Centres (Mississauga), Mississauga, Ontario
  - Oakville Trafalgar Memorial Hospital, Oakville, Ontario
  - James Cha, MD, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - CardioQuest Research Centre, Sarnia, Ontario
  - Niagara Health System - St. Catharines Site, St. Catharines, Ontario
  - Fadia El Boreky Medicine Professional Corporation, Waterloo, Ontario
  - ViaCar Recherches Cliniques Inc. (Brossard), Brossard, Quebec
  - Diex Recherche (Trois-Rivieres), Trois-Rivières, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
  - CIUSSS du Saguenay - Lac-Saint-Jean, Québec
  - CardioVasc HR Inc., Saint-Jean-sur-Richelieu
- Chile (6):
  - Enroll Spa, Santiago
  - CeCim - Centro de Estudios Clinicos e Investigacion Medica, Santiago
  - Centro de Investigación del Maule, Talca
  - Hospital Las Higueras, Talcahuano
  - CECMI Ltda, Temuco
  - CINVEC - Centro de Investigacion Clinica V Reg.,Vina del Mar, Viña del Mar
- China (66):
  - Beijing AnZhen Hospital, Capital Medical University, Beijing
  - Cardiovascular Institute and Fu Wai Hospital, Beijing
  - Jilin Province People's Hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - China-Japan Union Hospital of Jilin University, Changchun
  - Changde Second People's Hospital, Changde
  - Hunan Province People's Hospital (The First Affiliated Hospital of Hunan Normal University), Changsha
  - The Second Xiangya Hospital Of Central South University, Changsha
  - The Third Hospital of Changsha, Changsha
  - People's Hospital of Sichuan Province, Chengdu
  - Chenzhou No.1 people's Hospital, Chenzhou
  - Second Affiliated Hospital Chongqing Medical University, Chongqing
  - Chongqing Three Gorges Central Hospital, Chongqing
  - Affiliated Zhongshan Hospital of Dalian University, Dalian
  - Daqingshi People's Hospital, Daqing
  - People's Hospital of Deyang City, Deyang
  - The First People's Hospital of Foshan, Foshan
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Affiliated Panyu Central Hospital of Guangzhou Medical University, Guangzhou
  - Guizhou People's Hospital, Guiyang
  - Hainan General Hospital, Haikou
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - Jiangmen Central Hospital, Jiangmen
  - Center Hospital of Jinan, Jinan
  - Lanzhou University Second Hospital, Lanzhou
  - Linfen Central Hospital, Linfen
  - Luoyang Third People's Hospital, Luoyang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Jiangxi Province Integrated Tractional Chinese Medicine& Western Medicine Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - Nanjing Jiangning Hospital, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Nanyang First People's Hospital, Nanyang
  - Nanyang Second General Hospital, Nanyang
  - Ningbo Second Hospital, Ningbo
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Panjin Liao Oil Gem Flower Hospital, Panjin
  - Pingxiang People's Hospital, Pingxiang
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Tongren hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - People's Hospital of Liaoning Province, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Shanxi Bethune Hospital, Taiyuan
  - Shanxi Cardiovascular Hospital, Taiyuan
  - Taian City Central Hospital, Tai’an
  - Tianjin Union Medical Center Nankai University Affiliated Hospital, Tianjin
  - The 2nd Hospital of Tianjin Medical University, Tianjin
  - Hubei Province Zhongshan Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Shaanxi Provincial People's Hospital, Xi'an
  - Xinxiang Central Hospital, Xinxiang
  - The People's Hospital Of Xuancheng City, Xuancheng
  - The General Hospital of XZCMG (The Second Affiliated Hospital of Xuzhou Medical University), Xuzhou
  - The first People's Hosptal of Yinchuan, Yinchuan
  - Yueyang Central Hospital, Yueyang
  - Yuncheng Central Hospital, Yuncheng
  - The First Affiliated Hospital of Hebei North University, Zhangjiakoou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- Colombia (10):
  - Cardiomet CEQUIN S.A.S, Armenia
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
  - Corazon IPS S.A.S., Barranquilla
  - Fundacion Santa Fe de Bogota, Bogotá
  - Administradora Country S.A.S., Bogotá
  - Fundacion Hospital Infantil Universitario de San José, Bogotá
  - IPS Centro Medico Julián Coronel S.A., Cali
  - Centro de Diagnostico Cardiologico S.A.S., Cartagena
  - IPS médicos internistas de Caldas S.A.S., Manizales
  - T Y C Inversiones S.A.S Grupsalud, Santa Marta
- Czechia (19):
  - MUDr. Hana Burianova, Bílovec
  - Medicus Services Ltd., Brandýs nad Labem
  - Interni Ordinace s.r.o., Brandýs nad Labem
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - MUDr. Karel Kamenik s.r.o, Brno
  - MUDr. Jan Hubac s.r.o., Chrudim
  - EDUMED s.r.o., Jaroměř
  - MUDr Petra Maskova PhD, Litovel
  - KardioBusak s.r.o., Louny
  - InterKardioML s.r.o., Mariánské Lázně
  - MUDr. Zdenek Vomacka kardiologie a interna s.r.o., Olomouc
  - MUDr. Jan Kvasnicka CSc, Prague
  - Kardiologie Vinohrady s r o, Prague
  - Institute for Clinical and Experimental Medicine, Prague
  - University Hospital Motol, Prague
  - University Thomayer´s Hospital, Praha 4-Krc
  - Nemocnice Slany, Slaný
  - Kardiologicka ambulance MUDr. Ferkl s.r.o., Trutnov
  - Clinical Trials Services s.r.o, Uherské Hradiště
- Denmark (9):
  - Sygehus Sønderjylland Åbenrå, Aabenraa
  - Rigshospitalet Copenhagen, Copenhagen
  - Bispebjerg og Frederiksberg Hospital, Copenhagen NV
  - Amager-Hvidovre Hospital, Copenhagen S
  - Herlev and Gentofte Hospital, Herlev
  - Holbæk Sygehus, Holbæk
  - Hvidovre Hospital, Hvidovre
  - Sjællands Universitetshospital, Roskilde
  - Slagelse Sygehus, Slagelse
- Germany (27):
  - Klinikum am Plattenwald, Bad Friedrichshall
  - Universitätsklinikum Freiburg, Bad Krozingen
  - CIMS Studienzentrum Bamberg GmbH, Bamberg
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Velocity Clinical Research Germany GmbH, Berlin, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - GFO Kliniken Bonn, Betriebsstaette St. Marien, Bonn
  - Universitätsklinikum Bonn AöR, Bonn
  - SANA Kliniken Oberfranken Coburg GmbH, Coburg
  - Klinische Forschung Dresden GmbH, Dresden
  - Facharztzentrum Dresden-Neustadt Betriebsgesellschaft mbH, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Kardiopraxis Schirmer, Kaiserslautern
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Asklepios Klinik Langen-Seligenstadt GmbH, Langen
  - Klinikum der Stadt Ludwigshafen am Rhein GmbH, Ludwigshafen
  - Praxis Oedeme, Lüneburg
  - ze:ro Praxen MVZ fuer Nierenerkrankungen und Bluthochdruck GmbH Mannheim, Mannheim
  - Marienhaus Klinikum St. Elisabeth, Neuwied
  - Kardiologische Praxis Papenburg, Papenburg
  - Universitätsklinikum Regensburg, Regensburg
  - Gemeinschaftspraxis Dr. Josef Grosskopf und Dr. Wilma Grosskopf, Wallerfing
  - Kardiologische Praxis, Wermsdorf, Wermsdorf
  - Klinikum Worms gGmbH, Worms
- Hungary (15):
  - Belgyogyaszati es Kardiologiai Maganrendelo, Békéscsaba
  - Budai Irgalmasrendi Korhaz, Budapest
  - Obudai Egeszegugyi Centrum, Budapest
  - Belvaros-Lipotvaros Egeszsegugyi Szolgalat, Budapest
  - Gottsegen National Cardiovascular Center, Budapest
  - Semmelweis University, Budapest
  - Privat Doktor Egeszseguegyi Szolgaltato Zrt., Budapest
  - Zugloi Egeszsegugyi Szolgalat, Budapest
  - BKS Research Ltd, Hatvan
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - IPR Hungary Kft., Miskolc
  - TaNa Med Kft., Mosonmagyaróvár
  - Coromed-Smo Kft., Pécs
  - Tolna Varmegyei Balassa Janos Korhaz, Szekszárd
  - Belvarosi Egeszseghaz Kft., Zalaegerszeg
- India (15):
  - Kamal Nayan Bajaj Hospital, Aurangabad
  - Narayana Institute of Cardiac Sciences, Bangalore
  - S.P. Medical College & Associated Group of Hospitals, Bikaner
  - Tamil Nadu Government Multi Super Speciality Hospital TNGMSSH, Chennai
  - Apollo Hospital - Chennai, Chennai
  - Medanta-The Medicity, Gūrgaon
  - Lisie Hospital, Kochi
  - IPGMER and SSKM Hospital, Kolkata
  - Supe Heart & Diabetes Hospital & Research Centre, Nashik
  - Chopda Medicare and Research Centre Pvt Ltd, Nashik
  - Max Super Speciality Hospital, New Delhi
  - Indira Gandhi Institute of Medical Sciences, Patna
  - Nirmal Hospital, Surat
  - Unicare Heart Institute, Surat
  - King George Hospital, Visakhapatnam
- Italy (8):
  - Humanitas Gavazzeni, Bergamo
  - ASST Papa Giovanni XXIII, Bergamo
  - Az.Osp. Universitaria "Ospedali Riuniti", Foggia
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - Istituto Clinico Humanitas, Rozzano
- Japan (59):
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki-shi
  - Asahi General Hospital, Asahi-shi
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa-shi
  - Kyushu University Hospital, Fukuoka
  - Fukuokaken Saiseikai Futsukaichi Hospital, Fukuoka, Chikushino
  - Gunma University Hospital, Gunma, Maebashi
  - Minamino Cardiovascular Hospital, Hachioji-shi
  - National Hospital Organization Hamada Medical Center, Hamada-shi
  - JA-Shizuoka Enshu Hospital, Hamamatsu
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji-shi
  - Hiratsuka Kyosai Hospital, Hiratsuka-shi
  - Hitachi Ltd. Hitachinaka General Hospital, Hitachi-Naka
  - National Hospital Organization Kanazawa Medical Center, Ishikawa, Kanazawa
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni-shi
  - Tokushukai Shonan Kamakura General Hospital, Kamakura-shi
  - Tokushukai Hayama Heart Center, Kanagawa, Miura-gun
  - Mitoyo General Hospital, Kanonji-shi
  - Ibaraki Prefectural Central Hospital, Kasama-shi
  - Kasugai Municipal Hospital, Kasugai-shi
  - Saiseikai Kawaguchi Hospital, Kawaguchi-shi
  - St. Marianna University Hospital, Kawasaki-shi
  - Tokushukai Kishiwada Tokushukai Hospital, Kishiwada-shi
  - National Hospital Organization Kobe Medical Center, Kobe
  - Kumamoto University Hospital, Kumamoto
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Kure
  - Chibanishi General Hospital, Matsudo-shi
  - Shinshu University Hospital, Matsumoto-shi
  - Ehime Prefectural Central Hospital, Matsuyama
  - Matsuyama Shimin Hospital, Matsuyama
  - National Hospital Organization Tokyo Medical Center, Meguro-ku
  - Mito Saiseikai General Hospital, Mito
  - Tohoku University Hospital, Miyagi, Sendai
  - Sendai Cardiovascular Center, Miyagi, Sendai
  - Nagasaki Harbor Medical Center, Nagasaki, Nagasaki
  - Nagoya Kyoritsu Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Hokushin General Hospital, Nakano-shi
  - Nara Medical University Hospital, Nara, Kashihara
  - Juzenkai The Sakakibara Heart Institute of Okayama, Okayama, Okayama
  - Ome Municipal General Hospital, Ome-shi
  - Nagasaki Medical Center, Omura-shi
  - Osaka Metropolitan University Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Kosekai Iwatsuki-minami Hospital, Saitama, Saitama
  - Osaka Rosai Hospital, Sakaishi
  - Teine Keijinkai Hospital, Sapporo
  - NHO Sendai Medical Center, Sendai
  - NHO Kanmon Medical Center, Shimonoseki-shi
  - National Cerebral and Cardiovascular Center, Suita-shi
  - The University of Osaka Hospital, Suita-shi
  - Tachikawa Hospital, Tachikawa-shi
  - National Hospital Organization Takasaki General Medical Center, Takasaki-shi
  - NHO Minami Wakayama Medical Center, Tanabe-shi
  - Tokushima Prefectural Central Hospital, Tokushima
  - Tomakomai City Hospital, Tomakomai-shi
  - Toyota Memorial Hospital, Toyota-shi
  - NHO Shinshu Ueda Medical Center, Ueda-shi
  - Yokohama Sakae Kyosai Hospital, Yokohama
- Mexico (12):
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Centro Especializado de Investigación Medical Group Culiacan, Culiacán
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada S.C., Culiacán
  - Cardiologia Clinica e Intervencionista, Guadalajara
  - Proactive CR Mexico S.A. de C.V., Irapuato
  - Centro de Estudios de Alta Especialidad de Sinaloa CEAES, Mazatlán
  - Clinstile S.A. de C.V., México
  - Cardiolink Clin Trials S.C., Monterrey
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - Centro de Estudios Clinicos de Queretaro S.C, Querétaro
  - Centro de Investigacion Cardiovascular y Metabolica, Tijuana
  - CIMAB S.A. de C.V., Torreón
- Netherlands (7):
  - Jeroen Bosch Ziekenhuis-Hertogenbosch, 's-Hertogenbosch
  - Amsterdam University Medical Center, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Universitair Medisch Centrum Groningen, Groningen
  - Maastricht University Medisch Centrum, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - Isala Klinieken Stichting, Zwolle
- Poland (28):
  - Polsko-Amerykanskie Kliniki Serca, Bielsko-Biala
  - Centrum Medyczne Intercor Sp. z o.o., Bydgoszcz
  - Pratia Bydgoszcz Clinical Research Site, Bydgoszcz
  - NZOZ Medical Center KERmed, Bydgoszcz
  - Poradnia Kardiologiczna Jaroslaw Jurowiecki, Gdansk
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Specjalistyczna Praktyka Lekarska Ewa Mirek-Bryniarska, Krakow
  - Linden Sp. z o.o. sp.k., Krakow
  - Pratia MCM Krakow, Krakow
  - Beata Miklaszewicz & Dariusz Dabrowski Cardiamed Sp. j., Legnica
  - Santa SP. z o.o, Lodz
  - Velocity Nova Sp. z o.o., Lublin
  - Zanamed Medical Clinic Sp. z o.o., Lublin
  - Nzoz Heureka, Piaseczno
  - CBK Med Clinic SP Z O O, Płock
  - Centrum Medyczne Medyk, Rzeszów
  - Lukmed Lukasz Wozniak, Siedlce
  - Velocity Skierniewice Sp. z o.o, Skierniewice
  - Centrum Medyczne Pratia Poznan, Skórzewo
  - Velocity Staszow, Staszów
  - Sedimed Sp. z o.o., Szczecin
  - Balsammedica Sp. z o. o., Warsaw
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - ETG Warszawa, Warsaw
  - 4. Military Clinical Hospital with Polyclinic SP ZOZ, Wroclaw
  - Sedimed Sp. z o.o., Wroclaw
  - Velocity Nova Sp. z o.o., Zamość
  - Centrum Medyczne Serafin med, Żarów
- Romania (18):
  - Spitalul Judetean De Urgenta Dr. Constantin Opris Baia Mare, Baia Mare
  - Spitalul Clinic De Urgenta Prof Dr Agrippa Ionescu, Baloteşti
  - S.C.Centrul Medical Unirea S.R.L., Brasov
  - Spitalul Clinic Judetean de Urgenta Brasov, Brasov
  - Spitalul Judetean de Urgenta Braila, Brăila
  - Emergency University Hospital, Bucharest
  - Clinica Medicala Data Plus SRL, Bucharest
  - Cluj Napoca Clinical County Hospital, Cluj-Napoca
  - Spitalul Angiocare SRL, Cluj-Napoca
  - Emergency County Hospital Craiova, Craiova
  - Spitalul Clinic Judetean de Urgenta Bihor, Oradea
  - Sal Med Srl, Piteşti
  - U 2 Serv Com S.R.L., Suceava
  - Country Clinical Emergency Hospital, Targu-Mures, Târgu Mureş
  - Podoleanu G. Cristian-Gheorghe-Calin, Târgu Mureş
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
  - S.C Medicali's S.R.L, Timișoara
  - Timisoara Municipal Emergency Clinical Hospital, Timișoara
- Saudi Arabia (5):
  - King AbdulAziz University Hospital, Al Ahsa
  - King Fahad Specialist Hospital - Research Center, Dammam
  - Imam Abdulrahman bin Faisal University, Dammam
  - King Faisal Specialist Hospital and Research Center, Riyadh
  - King Fahad Medical City, Riyadh
- Serbia (9):
  - Clinical Center " Dr Dragisa Misovic Dedinje", Belgrade
  - University Clinical Center of Serbia, Belgrade
  - University Clinical Center of Kragujevac, Kragujevac
  - University Clinical Center Nis, Niš
  - Institute for Treatment and Rehabilitation, Niska Banja, Niška Banja
  - General Hospital Pancevo, Pančevo
  - General Hospital Sveti Luka, Smederevo
  - Institute of Cardiovascular Diseases of Vojvodine, Sremska Mitrovica
  - Health Centre Zajecar, Zaječar
- Slovakia (15):
  - Stredoslovensky Ustav Srdcovych A Cievnych Chorob A S, Banská Bystrica
  - Kardiointerna s r o, Banská Bystrica
  - Alian s.r.o., Bardejov
  - Cliniq s.r.o., Bratislava
  - Premedix Clinic, Bratislava
  - Nemocnica S Poliklinikou Brezno N.O., Brezno
  - Medical Group Kosice s.r.o, Košice
  - KARDIO R s r o, Košice
  - Cardio D&R s.r.o. Kosice, Košice
  - KARDIO 1 s.r.o., Lučenec
  - Kardiomed s.r.o., Lučenec
  - KVC Kardiovaskularne Centrum s.r.o., Martin
  - Cardiocenter Nitra, s.r.o, Nitra
  - Cardioamb s.r.o, Nové Zámky
  - Nemocnica AGEL Zvolen a.s., Zvolen
- South Korea (11):
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Yangsan Hospital, Busan
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (13):
  - Hospital Vall Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Virgen del Camino, Sanlúcar de Barrameda
  - Complexo Hospitalario Universitario De Santiago, Santiago de Compostela
  - Hospital Universitario De Torrejon, Torrejón de Ardoz
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Virgen de las Montañas, Villamartín
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang-Hua Christian Hospital, Taipei
- Turkey (Türkiye) (12):
  - Cukurova Universitesi Tip Fakultesi Gog. Hast. Anabilim Dali, Adana
  - Etlik City Hospital, Ankara
  - Ataturk Universitesi Tip Fakultesi, Erzurum
  - Osmangazi Uni Medical Faculty, Eskişehir
  - Gaziantep University Medical Faculty Sahinbey Educational Research Hospital, Gaziantep
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Medical Park Pendik Hospital, Istanbul
  - Dokuz Eylul University Faculty of Medicine, Izmir
  - Kutahya Health Science University, Kütahya
  - Inonu Uni. Med. Fac., Battalgazi, Malatya
  - Mersin University Medical Faculty, Mersin
  - Siyami Ersek Heart Hospital, Uskudar / Istanbul
- United Kingdom (5):
  - Southmead Hospital, Bristol
  - Royal Devon and Exeter Hospital, Wonford, Exeter
  - Calderdale Royal Hospital, Halifax
  - Northwick Park Hospital, Harrow
  - St Bartholomew's Hospital, London
- Vietnam (10):
  - Bach Mai hospital, Hanoi
  - Tam Anh General Hospital, Hanoi
  - Hanoi Heart Hospital, Hà Nội
  - Military Hospital 175, Ho Chi Minh City
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City
  - Tam Anh HCMC, Ho Chi Minh City
  - Thong Nhat Hospital HCMC, Ho Chi Minh City
  - Cho Ray Hospital, Ho Chi Minh City
  - University Medical Center HCMC, Ho Chi Minh City
  - Trung Vuong Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com